CLINICAL TRIAL: NCT06507319
Title: Comparative Evaluation Of Two Bone-Anchored Maxillary Molar Distalization Appliances: Direct Versus Indirect Anchorage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Zeyad Mahmoud, Dentist Zeyad Mahmoud, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Doctor Zeyad Mahmoud Ali
Record Dates: First submitted 2024-07-02; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Maxillary First Molar Distalization
Keywords: orthodontics; miniscrews; distalization; direct anchorage; indirect anchorage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct bone anchored pull distal slider (Experimental): The appliance will be cemented on the maxillary first molars and two miniscrews will be placed in their positions. The appliance will be activated by closed coil spring, which apply 300g force.
  Interventions: Device: Direct bone anchored pull distal slider
- Indirect bone anchored dual force distalizer. (Experimental): The appliance will be cemented on the teeth and two miniscrews will be placed in their positions. Activated by compressing the NiTi open coil spring from the buccal and palatal sides.
  Interventions: Device: Indirect bone anchored dual force distalizer.

INTERVENTIONS:
Device: Direct bone anchored pull distal slider — distalization from the palatal side only.
  Arms: Direct bone anchored pull distal slider
Device: Indirect bone anchored dual force distalizer. — distalization from the palatal and buccal sides.
  Arms: Indirect bone anchored dual force distalizer.

SUMMARY:
Aim of study: this study will be conducted for Comparative Evaluation Of Two Bone-Anchored Maxillary Molar Distalization Appliances: Direct Versus Indirect Anchorage.

Material and methods: The study will consist of two groups, each group has 10 Patients. The patients will be selected from the outpatient clinic of the orthodontic department at Mansoura University.

Patients will be divided into 2 groups, group 1 will be treated by direct bone anchored pull distal slider, and group 2 by indirect bone anchored dual force distalizer.

DETAILED DESCRIPTION:
Aim of study:

this study will be conducted for Comparative Evaluation Of Two Bone-Anchored Maxillary Molar Distalization Appliances: Direct Versus Indirect Anchorage.

Participant and eligibility criteria:

The study will consist of two groups, each group has 10 Patients. The patients will be selected from the outpatient clinic of the orthodontic department at Mansoura University. pretreatment records will be taken including: intraoral and extraoral photographs, study models, panoramic radiographs, and lateral cephalometric radiographs.

Intervention:

written and informed consents will be taken from the patients.

Group 1:

* Two metal bands will be chosen and fitted on the maxillary first molars.
* Rubber base impression material will be taken with bands in place.
* Two metal bands will be placed in their relative positions in the impression and then poured up with stone.
* Send it to the LAB for appliance fabrication.
* At delivery day, the appliance will be cemented on the maxillary first molars by glass ionomer luting cement and two miniscrews will be placed in their positions.
* The appliance will be activated by closed coil spring, which apply 300g force. Patients will be monitored every 3 weeks.

Group 2:

* Four metal bands ( two for maxillary first premolars and two for maxillary first molars ) will be chosen and fitted on the teeth.
* Rubber base impression material will be taken with bands in place.
* Four metal bands will be placed in their relative positions in the impression and then poured up with stone.
* Send it to the LAB for appliance fabrication.
* At delivery day, the appliance will be cemented on the teeth by glass ionomer luting cement and two miniscrews will be placed in their positions, and activated by compressing the NiTi open coil spring, which apply 300g force. Patients will be monitored every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Dental class II.
* No or mild to moderate maxillary teeth crowding.
* Erupted or partially erupted maxillary second molars.
* No previous orthodontic therapy.
* Absence or minimum crowding in the mandibular arch.
* Good oral hygiene.

Exclusion Criteria:

* Dental class I, III
* severe maxillary teeth crowding.
* Extracted or badly decayed maxillary first molars.
* Previous orthodontic therapy.
* Severe crowding in the mandibular arch.
* Bad oral hygiene.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Anteroposterior skeletal measurements | 8 months
  From the lateral cephalometric, the maxillary and mandibular sagittal positions will be measured according to the SN plane, before and after distalization.
Vertical skeletal measurements | 8 months
  From the lateral cephalometric, mandibular plane angle according to the SN plane and Frankfort horizontal plane, will be measured before and after distalization.
Dental angular measurements | 8 months
  From the lateral cephalometric, the angle between teeth (maxillary central incisor, first premolar, second premolar, first molar) and the SN plane will be measured before and after distalization to measure the amount of tipping.
Amount of distalization | 8 months
  From the lateral cephalometric, the distance between teeth (maxillary central incisor, first premolar, second premolar, first molar) and the pterygoid vertical (PTV) plane will be measured before and after distalization to calculate the amount of distalization in mm.
Amount of intrusion | 8months
  From the lateral cephalometric, the distance between teeth (maxillary central incisor, first premolar, second premolar, first molar) and the palatal plane (PP) will be measured before and after distalization to calculate the amount of intrusion in mm.
  .
Amount of expansion | 8 months
  From the study model, the maxillary inter-canine, inter-first premolar, inter-second premolar, inter-first molar, and inter-second molar widths will be measured before and after distalization to calculate the amount of expansion in mm.
Amount of rotation | 8 months
  From the study model, the angle between buccopalatal axis of teeth (maxillary first premolar, second premolar, first molar) and the midpalatal suture will be measured before and after distalization to calculate the amount of rotation.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No